CLINICAL TRIAL: NCT03079271
Title: An Open Label Comparing the Short Term Efficacy of Lacrisert
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Virginia Eye Consultants (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: VEC-LAC001
Record Dates: First submitted 2016-11-23; First posted 2017-03-14 (Actual); Last update posted 2017-03-14 (Actual); Status verified 2017-03

CONDITIONS: Dry Eye
MeSH Terms: conditions — Dry Eye Syndromes | interventions — hydroxypropylcellulose

ARMS (1):
- open label (Other)
  Interventions: Drug: Lacrisert, 5 Mg Ophthalmic Insert

INTERVENTIONS:
Drug: Lacrisert, 5 Mg Ophthalmic Insert

SUMMARY:
To evaluate the short term effects of LACRISERT®. upon fluorescein corneal staining, tear osmolarity and surface topography in human subjects with dry eye disease.

ELIGIBILITY:
Inclusion Criteria:

-Has Dry Eye disease indicated by a staining score of ≥ 4 and Speed score of >6

Exclusion Criteria:

* Concurrent involvement in any other clinical trial
* Anticipated contact lens wear during the study and 14hours prior to Day -History of corneal transplant
* Active ocular infection, uveitis or non-KCS inflammation
* History of recurrent herpes keratitis or active disease within the last six months
* Topical ophthalmic medications during the study
* Temporary collagen punctal plugs within one week prior to study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2016-11; Primary Completion 2017-06 (Estimated); Study Completion 2017-12 (Estimated)

PRIMARY OUTCOMES:
Dry Eye disease measured by OSDI questionnaire | 10 days
Dry eye disease measured by Corneal Staining | 10 days
Dry eye disease measured by topographic results | 10 days

CONTACTS AND LOCATIONS:
Locations (1):
- Virginia Eye Consultants, Norfolk, Virginia, United States